CLINICAL TRIAL: NCT02685293
Title: A Randomized, Phase IIIb, Two-period , Double-blind, Two-treatment, Chronic-dosing (7 Days), Single-center Crossover Study to Evaluate the Treatment Effect of PT003 on Cardiovascular Hemodynamics in Subjects With Moderate to Severe Chronic Obstructive Pulmonary Disease, Compared With Placebo
Brief Title: Study to Evaluate the Treatment Effect of PT003 on Cardiovascular Hemodynamics in Subjects With Moderate to Severe COPD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PT003017
Record Dates: First submitted 2016-01-28; First posted 2016-02-18 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GFF MDI (PT003) (Experimental): Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI)
  Interventions: Drug: GFF MDI (PT003)
- Placebo MDI (Placebo Comparator): Placebo Metered Dose Inhaler (MDI) for Glycopyrronium and Formoterol Fumarate Inhalation Aerosol
  Interventions: Drug: Placebo MDI

INTERVENTIONS:
Drug: GFF MDI (PT003) — Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI)
  Arms: GFF MDI (PT003)
Drug: Placebo MDI — Placebo Metered Dose Inhaler (MDI) for Glycopyrronium and Formoterol Fumarate Inhalation Aerosol
  Arms: Placebo MDI

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single-center, chronic-dosing (7 days), two-period, two-treatment, cross-over study to evaluate the treatment effect of PT003 compared with that of Placebo MDI on Cardiovascular Hemodynamics following chronic-dosing (7 days) in subjects with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* At least 40 years of age and no older than 80 at Visit 1.
* Women of non-child bearing potential,or negative serum pregnancy test at Screening, and agrees to acceptable contraceptive methods used consistently and correctly from Screening until 14 days after final visit
* Evidence of lung hyperinflation
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking.
* Pre- and Post-bronchodilator FEV1/FVC ratio must be <0.70
* Post-bronchodilator FEV1 must be ≥30% to <65% predicted normal value, calculated using NHANES III reference equations.

Exclusion Criteria:

* Significant diseases or conditions other than COPD which, in the opinion of the Investigator, may put the patient at risk
* Women who are pregnant or lactating or are planning to become pregnant during the course of the study
* Subjects, who in the opinion of the Investigator, have a current diagnosis of asthma or other active pulmonary disease
* Subjects who have been hospitalized due to poorly controlled COPD within 3 months prior to Screening
* Subjects who have poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to Screening or during the Screening Period
* Subjects who have clinically significant uncontrolled hypertension.
* Subjects with symptomatic prostatic hypertrophy that is clinically significant and not adequately controlled with appropriate therapy, in the opinion of the Investigator.
* Subjects with bladder neck obstruction or urinary retention that is clinically significant in the opinion of the Investigator.
* Subjects with a calculated creatinine clearance ≤30 mL/minute using Chronic Kidney Disease Epidemiology Collaboration. (CKD-EPI) formula at Screening and on repeat testing prior to Visit 2.
* Subjects with abnormal liver function tests defined as AST, ALT, or total bilirubin ≥ 1.5 times upper limit of normal at Screening and on repeat testing prior to Visit 2
* Subjects who have cancer that has not been in complete remission for at least five years.
* Subjects with a diagnosis of glaucoma, who in the opinion of the Investigator, have not been adequately treated.
* Subjects with a clinically significant ECG
* Subjects who were previously enrolled in any previous PT001, PT003, or PT005 study conducted or sponsored by Pearl.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, MD, Study Chair — Pearl Therapeutics
Locations (1):
- Research Site, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
AstraZeneca's policy is to share data with researchers if the request is in scope of our policy. The policy and additional information can be found on astrazenecaclinicaltrials.com.

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4146&filename=PT003017_CSP_V3_Redacted_coverpage_PDFA.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with moderate to severe chronic obstructive pulmonary disease (COPD) were enrolled into this 2-period, 2-treatment, crossover study from 09 December 2016. The study was terminated early on 20 June 2018.
Pre-assignment Details: Subjects were randomly assigned, in a 1:1 ratio, to receive either Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI) then Placebo MDI or Placebo MDI then GFF MDI in two 7-day treatment periods, separated by a washout period of between 7 and 21 days.
Groups:
- GFF MDI, Then Placebo MDI: Subjects first received GFF MDI (PT003) 14.4/9.6 micrograms (μg) as 2 inhalations twice daily (BID) for 7 days in treatment period 1. After a washout period, subjects then received Placebo MDI as 2 inhalations BID for 7 days in treatment period 2.
- Placebo MDI, Then GFF MDI: Subjects first received Placebo MDI as 2 inhalations BID for 7 days in treatment period 1. After a washout period, subjects then received GFF MDI 14.4/9.6 μg as 2 inhalations BID for 7 days in treatment period 2.
Period: Treatment Period 1
Arm/Group | GFF MDI, Then Placebo MDI | Placebo MDI, Then GFF MDI
Started | 1 | 3
Completed | 1 | 3
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | GFF MDI, Then Placebo MDI | Placebo MDI, Then GFF MDI
Started | 1 | 3
Completed | 1 | 3
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | GFF MDI, Then Placebo MDI | Placebo MDI, Then GFF MDI
Started | 1 | 3
Completed | 1 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Subjects: All subjects randomized to receive treatment.
Arm/Group | All Randomized Subjects
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Right Ventricular End Diastolic Volume Index (RVEDVi) at 2-3 Hours Post-dose on Day 8
Description: Assessment of right ventricular (RV) volume was performed using magnetic resonance imaging (MRI) using RV end diastolic volume (RVEDV), 2-3 hours after dosing on Day 8 of each treatment period. RVEDV was normalized to body surface area (BSA) to provide the indexed counterpart (RVEDVi). Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: cm^3/m^2
Groups:
- GFF MDI: GFF MDI (PT003) 14.4/9.6 μg was administered as 2 inhalations BID for 7 days in either treatment period 1 or treatment period 2.
- Placebo MDI: Placebo MDI was administered as 2 inhalations BID for 7 days in either treatment period 1 or treatment period 2.
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 4 | 4
cm^3/m^2 | 6.10 (7.69) | -7.93 (8.64)

2. Secondary Outcome: Change From Baseline in Aortic Left Ventricular Stroke Volume (LVSV) at 2-3 Hours Post-dose on Day 8
Description: Assessment of LVSV was performed using MRI, 2-3 hours after dosing on Day 8 of each treatment period. Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 4 | 4
cm^3 | 8.40 (14.14) | 2.88 (12.61)

3. Secondary Outcome: Change From Baseline in Right Ventricular Stroke Volume (RVSV) at 2-3 Hours Post-dose on Day 8
Description: Assessment of RVSV, phase contrast from pulmonic valve, was performed using MRI, 2-3 hours after dosing on Day 8 of each treatment period. Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 4 | 4
cm^3 | 8.38 (12.74) | 2.83 (12.40)

4. Secondary Outcome: Change From Baseline in Pulmonary Artery Velocity at 2-3 Hours Post-dose on Day 8
Description: Assessment of Pulmonary Artery Velocity was performed using MRI, 2-3 hours after dosing on Day 8 of each treatment period. Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: cm/second
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 4 | 4
cm/second | 0.91 (1.67) | -0.15 (1.43)

5. Secondary Outcome: Change From Baseline in Left Ventricular End Diastolic Volume Index (LVEDVi) at 2-3 Hours Post-dose on Day 8
Description: Assessment of left ventricular (LV) volume was performed using MRI using LV end diastolic volume (LVEDV), 2-3 hours after dosing of Day 8 of each treatment period. LVEDV was normalized to BSA to provide the indexed counterpart (LVEDVi). Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: cm^3/m^2
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 4 | 4
cm^3/m^2 | 6.95 (6.47) | -1.77 (6.44)

6. Secondary Outcome: Change From Baseline in Cardiac Output at 2-3 Hours Post-dose on Day 8
Description: Assessment of cardiac output was performed using MRI, 2-3 hours after dosing on Day 8 of each treatment period. Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 4 | 4
Liters/minute | 0.95 (0.80) | 0.38 (1.17)

7. Secondary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR) at 30 and 60 Minutes Post-dose on Day 8
Description: Assessment of PVR was performed by impedance cardiography at 30 and 60 minutes after dosing on Day 8 of each treatment period. Baseline for was defined as the average of the subject values obtained pre-dose on Day 1 of each treatment period.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: Due to early termination of the study, data for this endpoint were not collected.
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Pulmonary Artery/Aortic Diameter Ratio (PA:A) at 2-3 Hours Post-dose on Day 8
Description: Assessment of PA:A was performed using MRI, 2-3 hours after dosing on Day 8 of each treatment period. Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 4 | 4
ratio | -0.03 (0.15) | -0.04 (0.21)

9. Secondary Outcome: Change From Baseline in Left Atrial End Diastolic Volume (LAEDV) at 2-3 Hours Post-dose on Day 8
Description: Assessment of LAEDV was performed using MRI, 2-3 hours after dosing on Day 8 of each treatment period. Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: Due to early termination of the study, data for this endpoint were not collected.
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Left Atrial End Systolic Volume (LAESV) at 2-3 Hours Post-dose on Day 8
Description: Assessment of LAESV was performed using MRI, 2-3 hours after dosing on Day 8 of each treatment period. Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: Due to early termination of the study, data for this endpoint were not collected.
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Left Atrial Ejection Fraction (LAEF) at 2-3 Hours Post-dose on Day 8
Description: Assessment of LAEF was performed using MRI, 2-3 hours after dosing on Day 8 of each treatment period. Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: Due to early termination of the study, data for this endpoint were not collected.
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in Left Ventricular End Systolic Volume Index (LVESVi) at 2-3 Hours Post-dose on Day 8
Description: Assessment of LV volume was performed using MRI using LV end systolic volume (LVESV), 2-3 hours after dosing on Day 8 of each treatment period. LVESV was normalized to BSA to provide the indexed counterpart (LVESVi). Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: cm^3/m^2
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 4 | 4
cm^3/m^2 | 2.68 (2.56) | -3.18 (2.06)

13. Secondary Outcome: Change From Baseline in Right Ventricular End Systolic Volume Index (RVESVi) at 2-3 Hours Post-dose on Day 8
Description: Assessment of RV volume was performed using MRI using RV end systolic volume (RVESV), 2-3 hours after dosing on Day 8 of each treatment period. RVESV was normalized to BSA to provide the indexed counterpart (RVESVi). Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: cm^3/m^2
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 4 | 4
cm^3/m^2 | 1.92 (5.95) | -9.23 (4.64)

14. Secondary Outcome: Change From Baseline in Pulsatility Index Aorta (PIAo) at 2-3 Hours Post-dose on Day 8
Description: Assessment of PIAo was performed using MRI, 2-3 hours after dosing on Day 8 of each treatment period. Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 4 | 4
percent | -0.63 (13.45) | -0.37 (4.07)

15. Secondary Outcome: Change From Baseline in Pulmonary Artery Pulsatility Index (PAPi) at 2-3 Hours Post-dose on Day 8
Description: Assessment of PAPi was performed using MRI, 2-3 hours after dosing on Day 8 of each treatment period. Baseline was defined as the pre-dose value on Day 1 of treatment period 1.
Time Frame: Baseline and Day 8 of either treatment period 1 or 2, as applicable.
Population: All randomized subjects.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | GFF MDI | Placebo MDI
Number analyzed (Participants) | 4 | 4
percent | 3.60 (10.86) | -4.95 (19.54)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from screening, throughout the treatment periods until the follow-up visit 14±2 days from the last study treatment administration. Overall timeframe of up to a maximum of 12 weeks.
Groups:
- Placebo: Placebo MDI was administered as 2 inhalations BID for 7 days in either treatment period 1 or treatment period 2.
Arm/Group | GFF MDI | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI (N=4) | Placebo (N=4)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early on 20 June 2018 as target enrollment numbers were not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT02685293/Prot_SAP_000.pdf